CLINICAL TRIAL: NCT01052896
Title: Gabapentin in Functional Dyspepsia Refractory to Proton Pump Inhibition
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit subjects - unworkable
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWH20090188H; WS499026 (Other Grant/Funding Number: Pfizer Pharmaceuticals)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Functional Dyspepsia
Keywords: Dyspepsia; Functional
MeSH Terms: conditions — Dyspepsia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Half of the 100 patients enrolled will be placed on Gabapentin therapy to determine if they have improved dyspepsia symptoms.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Half of the 100 patients will be placed on placebo look-alike of the gabapentin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — 300mg po TID
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Look-alike of gabapentin 300mg given po tid
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of gabapentin on symptom control in patients with defined functional dyspepsia refractory to conventional proton pump inhibitor therapy and to compare these effects to that of placebo.

DETAILED DESCRIPTION:
In this pilot study we hypothesize that the patients on gabapentin will have an increase in the adequacy of dyspepsia symptom control at two months as well as improvement in dyspepsia symptom index scores which are a surrogate of quality of life measures, when compared to placebo.

While functional dyspepsia is divided into four subtypes most studies have grouped all four as 'functional dyspepsia' and treated them as one. Proton pump inhibition may benefit those with epigastric pain or burning but typically not those with post-prandial fullness or early satiety. (Tack et al). Those patients with symptoms refractory to proton pump inhibition might benefit from a medication that modifies visceral hypersensitivity such as gabapentin. It is possible that by modifying their pain syndrome we can decrease the need for follow-up appointments and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be included in this study are adults (age >18 years) with defined functional dyspepsia per the ROME III criteria with a negative EGD who are on proton pump inhibitor therapy yet still have a sense of inadequate symptom control.

Exclusion Criteria:

* Patients excluded will be women of childbearing age who refuse to have a baseline pregnancy test and/or who refuse to prevent pregnancy during the trial period. Exclusion criteria will also include anyone with a history of adverse effect or allergy to gabapentin. Finally, any patient undergoing hemodialysis or with a history of creatinine chronically greater than 1.5 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03 (Estimated); Primary Completion 2011-03 (Estimated); Study Completion 2012-08-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the adequacy of symptom control during the last week of the study. | 2 months

SECONDARY OUTCOMES:
Secondary outcomes equate dyspepsia symptoms with quality of life. The Nepean Dyspepsia Index scores patients on five categories while the Global Overall Symptom Scale measures the severity of dyspepsia on a 1-7 scale. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Molloy, MD, Principal Investigator — Gastroenterology Division - SAMMC
Locations (2):
- United States (2):
  - San Antonio Military Medical Center - North, San Antonio, Texas
  - San Antonio Military Medical Center - South, San Antonio, Texas